CLINICAL TRIAL: NCT03550521
Title: A Mixed Methods Investigation of Brief Mindfulness Training and Self-injury Attentional Bias Among Self-injuring Adolescents
Brief Title: Interrupting Self-Harm Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB_00108383
Record Dates: First submitted 2018-05-09; First posted 2018-06-08 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Nonsuicidal Self-injury
MeSH Terms: conditions — Self-Injurious Behavior | interventions — Mindfulness

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness condition (Experimental): The brief mindfulness induction will be modeled after basic mindfulness skills commonly used in mindfulness-based interventions and tailored to target distressing thoughts and feelings.
  Interventions: Behavioral: Mindfulness
- Control condition (No Intervention): Participants assigned to the control task will be instructed to "let your mind wander freely without trying to focus on anything in particular."

INTERVENTIONS:
Behavioral: Mindfulness — Participants will be instructed to focus on the sensations of breathing. Subsequently, whenever their minds wander to distressing thoughts or emotions, they will be instructed to acknowledge those thoughts or emotions, and then bring their attention back to the sensations of breathing.
  Arms: Mindfulness condition

SUMMARY:
My study will employ a convergent mixed methods two-arm parallel randomized controlled design. The qualitative strand will primarily rely on semi-structured interview procedures to answer the following questions: (1) How do adolescents perceive and experience the phenomenon of nonsuicidal self-injury (NSSI)? (2) What do adolescents believe needs to be done to address NSSI? The quantitative strand will primarily rely on clinical interview data, self-report measures, and an experimental task protocol to answer the following question: What is the impact of a brief mindfulness induction (versus a control condition) on self-injury attentional bias among self-injuring adolescents?

ELIGIBILITY:
Inclusion Criteria:

* To be included in the study, a participant must be: 1) at least 12 years old and no more than 18 years old, 2) able to understand and communicate in English, 3) willing and able to participate in all study procedures, and 4) currently engaging in nonsuicidal self-injury OR have a history of nonsuicidal self-injury.

Exclusion Criteria:

* Individuals will be excluded from the study if they are experiencing a suicidal crisis at the time of the study procedures (e.g., they endorse suicidal ideation, planning, and intent as determined by the Mini International Neuropsychiatric Interview 7.0) and require crisis intervention or hospitalization.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Change in self-injury attentional bias as measured by a Dot Probe Paradigm | The Dot Probe Paradigm will be administered immediately preceding the mindfulness or control conditions and immediately following the mindfulness or control conditions
  Attentional bias (AB) refers to the allocation of attentional resources to specific aspects of environmental stimuli

CONTACTS AND LOCATIONS:
Overall Officials: Michael R Riquino, MSW, Principal Investigator — University of Utah College of Social Work
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Interventions for self-harm in children and adolescents. Cochrane Database Syst Rev. 2021 Mar 7;3(3):CD013667. doi: 10.1002/14651858.CD013667.pub2. PMID 33677832